CLINICAL TRIAL: NCT04828304
Title: PLASOMA Ultimate Safety & Efficacy Study
Acronym: PULSE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Plasmacure (Industry)
Collaborators: Diabetes Fonds (Other); Pathology and Medical Microbiology (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PULSE study
Record Dates: First submitted 2021-03-24; First posted 2021-04-02 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-05

CONDITIONS: Diabetic Foot Ulcer; Venous Leg Ulcer; Pressure Ulcer; Burn Wound; Skin Graft; Infected Surgical Wound; Skin Flap
MeSH Terms: conditions — Diabetic Foot; Varicose Ulcer; Pressure Ulcer; Burns; Surgical Wound Infection

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- control group (No Intervention): Standard of care
- treatment group (Experimental): Standard of care + PLASOMA treatment
  Interventions: Device: PLASOMA

INTERVENTIONS:
Device: PLASOMA — Treatment with cold plasma device
  Arms: treatment group

SUMMARY:
The purpose of the PULSE study are the followingL

A.To perform post market clinical follow up (PMCF) on safety and efficacy:

1. Safety: To confirm transient short-terms side effects and verify long-term/outstanding risks.
2. Efficacy: To confirm the performance of PLASOMA, i.e. the beneficial effect on bacterial load. B. Determine the effect of PLASOMA on wound surface area.

A secondary purpose is to examine the beneficial effects of PLASOMA on wound healing and to perform a health technology assessment (HTA).

This clinical study will be an open label two-armed randomized controlled trial (RCT), performed at at least three sites (multi-center) in the Netherlands.

The two arms are:

1. Control group: Standard wound care for 12 weeks or until healing, whichever occurs first;
2. Treatment group: Standard wound care + PLASOMA treatment for 12 weeks or until healing, whichever occurs first.

The frequency of PLASOMA treatment will be determined by the treating (para)medical professional based on the number of visits they would schedule for the standard wound care at the study site.

For all study subjects, the treatment frequency will be at least once per week (in order to have enough treatments for safety evaluation) and should not exceed once per day.

Follow up (FU) will be performed at three timepoints for both arms:

* FU1: 2 weeks after end treatment period
* FU2: 12 weeks after end treatment period
* FU3: 12 months after start treatment.

ELIGIBILITY:
Inclusion criteria:

INCL1: have a slow-healing or non-healing ulcer consisting of, but not limited to:

* diabetic ulcers (Wagner-Meggitt classification system/ University of Texas classification system: grades 1-3)
* venous ulcers
* pressure ulcers (international NPUAP/EPUAP classification system: categories/stages II-IV)
* burn wounds (second and third degree)
* skin grafts and flaps
* infected post-surgical ulcers. Standard wound care has not resulted in sufficient healing after at least two weeks (including first line care) (Ref 25, Ref 26).

Note: There is no upper limit for the duration that the wound exists. In case a subject has multiple wounds that meet the in- and exclusion criteria, the wound with the longest duration will be chosen for the study.

INCL2: have a wound with a minimum wound surface area of 0.5 cm2 and a maximum diameter of 4.5 cm (~16 cm2 wound surface area for circular wounds).

INCL3: have a minimum age of 18 years old.

INCL4: for home care treatments only: have a grounded wall socket available for connection of PLASOMA.

Exclusion criteria:

EXCL1: the subject has one or more of the following contraindications for PLASOMA:

* the wound is very exudative, i.e. wounds in which moisture is visible again within a few minutes after patting dry.
* any implanted active electronic device, such as a pacemaker, is present.
* an electronic medical device is attached to the body, including electronic life support equipment, hearing aids, glucose sensors and insulin pumps. If the sole purpose of the medical device is monitoring, the subject is not excluded, but it should be noted that use of PLASOMA together with such devices has not been tested and may lead to erroneous operation of the attached device during PLASOMA treatment.
* Note: no exclusion if electronic medical device will be detached during PLASOMA treatment.
* a metal implant (including a stent) is present in the treatment area, i.e. the area between pad and electrode.
* a conductive connection from outside to inside the body at or near the heart is present, e.g. a catheter with electrolyte fluid.
* the subject has epilepsy
* the subject is pregnant
* the to-be-treated wound is located on the torso above the navel

EXCL2: the subject has any known malignant wound degeneration.

EXCL3: the subject receives treatment with immunosuppressive agents or oral corticosteroids; no exclusion if subject has received a stable dose for at least 2 months and the oral corticosteroid dose does not exceed 7.5 mg/day prednisone or equivalent.

EXCL4: the subject is receiving or likely to receive advanced wound therapies - such as negative pressure therapy, hyperbaric oxygen therapy, biologicals (e.g. skin substitutes, growth factors), electrophysical therapy - until FU1 for the to be-treated wound. Advanced wound dressings are not excluded.

EXCL5: the subject participates in another study which is likely to compromise the outcome of the PULSE study or the feasibility of the subject fulfilling the PULSE study.

EXCL6: the subject is unable to provide consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2021-05-26 (Actual); Primary Completion 2024-12-16 (Actual); Study Completion 2024-12-16 (Actual)

PRIMARY OUTCOMES:
Safety PLASOMA - device related SAEs | 12 months
  device related SAEs
Efficacy PLASOMA - bacterial load reduction - Staphylococcus aureus | once at week 1 (wound swab directly before and after first PLASOMA treatment)
  Reduction in number of S. aureus colonies, using wound swab and quantitative analysis
Efficacy PLASOMA - wound surface area reduction | 12 weeks
  Wound surface area reduction

SECONDARY OUTCOMES:
Safety PLASOMA - all AEs | 12 months
  Safety reporting
Safety PLASOMA - wound appearance | 24 weeks
  wound appearance
Efficacy PLASOMA - Bacterial load reduction | once at week 1 (wound swab directly before and after first PLASOMA treatment)
  Bacterial load reduction (total load and Pseudomonas aeruginosa), using wound swab and semi-quantitative analysis
Efficacy PLASOMA- wound healing | 12 weeks
  Wound healing - wound surface area reduction - wound volume reduction - time to healing
Efficacy PLASOMA - Quality of Life | 14 weeks
  Quality of Life, using RAND-36 questionnaire
Efficacy PLASOMA - Quality of Life | 14 weeks
  Quality of Life, using Wound-QoL questionnaire
Efficacy PLASOMA - Ulcer recurrence | 12 months
  Ulcer recurrence
Efficacy PLASOMA - wound infection | 12 weeks
  wound infection (clinical classification)
Efficacy PLASOMA - wound pain | 12 weeks
  wound pain (0-10 numerical rating scale)
Health Technology Assessment PLASOMA | 12 weeks
  resource usage PLASOMA
Patient acceptability | 12 weeks
  Patient acceptability (subjects will be asked if they are happy with the PLASOMA treatment)

CONTACTS AND LOCATIONS:
Overall Officials: Koen Lim, Study Director — Plasmacure
Locations (6):
- Netherlands (6):
  - Groene Hart Ziekenhuis, Gouda
  - Alrijne Ziekenhuis, Leiderdorp
  - Sint Antonius Ziekenhuis, Nieuwegein
  - radboud Universitair Medisch Centrum, Nijmegen
  - Expertisecentrum Wondzorg (EcW), Oosterhout
  - Maxima Medisch Centrum (MMC), Veldhoven